CLINICAL TRIAL: NCT02960269
Title: Interprofessional Management of Chronic Back Pain in Rural and Remote Setting: Use of Telehealth vs. Secure Laptop-based Videoconferencing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Kelsey Trail Health Region (Other)
Responsible Party: Principal Investigator, Brenna Bath, Assistant Professor, University of Saskatchewan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Bio16-49
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Back Pain Lower Back Chronic
Keywords: rural health; telehealth; physiotherapy; interprofessional

ARMS (1):
- Telehealth team assessment (Experimental): Team assessment for back pain with nurse practitioner and physical therapist via telehealth
  Interventions: Other: interprofessional back pain assessment

INTERVENTIONS:
Other: interprofessional back pain assessment — team assessment and education with urban physical therapist and rural nurse practitioner via telehealth

SUMMARY:
This pilot study will evaluate the impact and overall experience of an interprofessional chronic low back pain patient care approach for people in rural and remote areas using Telehealth technology compared to secure laptop based videoconferencing (Vidyo).

DETAILED DESCRIPTION:
People with chronic low back pain will be recruited to participate in a team assessment with a local rural nurse practitioner and an-urban based physiotherapist linking through telehealth. The assessment will include a detailed history, physical examination and jointly-delivered education and recommendations for further community-based management. Pre and post measures of self-reported pain, back-specific function, quality of life, and satisfaction will be completed 2-4 weeks after the assessment. Comparison of short-term outcomes will be made with a group of participants from another study using the a different telehealth technology (secure laptop based videoconferencing) same inclusion criteria, measures and health care providers (Clin Trials.gov NCT02225535). The health care providers will be interviewed to get feedback on their preference and experience using the different type of telehealth technology.

ELIGIBILITY:
Inclusion Criteria:

chronic low back pain localized below costal margins and above gluteal folds and/or related leg pain, which is bad enough to limit their usual activities or daily routine and has been present for at least 3 months

Exclusion Criteria:

* People with: third party payer insurance (i.e.worker's compensation board) for their back related complaints, with primarily neck or thoracic pain, and/ or with language, reading or comprehension barriers that would limit their ability to adequately complete the required study paperwork will be excluded from participating in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-11; Primary Completion 2017-03 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Patient experience with telehealth | 2-4 weeks after assessment
Pain | 2-4 weeks after assessment
  Numeric Pain Rating Scale
Back-specific function | 2-4 weeks after assessment
  Modified Oswestry Disability Index
Participant satisfaction | 2-4 weeks after assessment
  Modified VSQ-9

SECONDARY OUTCOMES:
Health care provider experience | within 2 weeks of completion of all assessments
  experience with telehealth technology

CONTACTS AND LOCATIONS:
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada